CLINICAL TRIAL: NCT01659242
Title: Leflunomide Versus Sulfasalazine/Methotrexate in Rheumatoid Arthritis Patients With Active Disease Despite Methotrexate: an Ultrasound and Magnetic Resonance Imaging Study
Brief Title: Leflunomide Versus Sulfasalazine/Methotrexate in Rheumatoid Arthritis:an Ultrasound/Magnetic Resonance Imaging Study
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: YK 01-2012
Record Dates: First submitted 2012-08-03; First posted 2012-08-07 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis; Ultrasound; Magnetic Resonance Imaging
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Methotrexate; Sulfasalazine; Leflunomide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Methotrexate plus sulfasalazine (Active Comparator): ARM 1(Methotrexate(MTX) plus Sulfasalazine(SSZ))
  SSZ:Oral form, 2g/day, with escalation regime starting from 1g/day for the first week and increase to 1.5g/day in the next week and increasing to 2g/day by the third week. Total treatment period is 16 weeks. After reaching 2g/day, if patients conditions warrants (and no contraindication), SSZ may be increased at 0.5g per clinic visit) up to a maximum of 3g/day.
  MTX:Kept at the highest optimal dose.
  Interventions: Drug: Methotrexate plus sulfasalazine
- Leflunomide (Active Comparator): ARM 2:Leflunomide(LEF)
  LEF: Oral form, 20mg every other day for first 2 weeks then increasing to 20mg per day by the third week. Total treatment period is 16 weeks.
  Methotrexate:Off
  Interventions: Drug: Leflunomide

INTERVENTIONS:
Drug: Methotrexate plus sulfasalazine — ARM 1(Methotrexate(MTX) plus Sulfasalazine(SSZ))
  SSZ:Oral form, 2g/day, with escalation regime starting from 1g/day for the first week and increase to 1.5g/day in the next week and increasing to 2g/day by the third week. Total treatment period is 16 weeks. After reaching 2g/day, if patients conditions warrants (and no contraindication), SSZ may be increased at 0.5g per clinic visit) up to a maximum of 3g/day.
  MTX:Kept at the highest optimal dose.
  Arms: Methotrexate plus sulfasalazine
Drug: Leflunomide — ARM 2:Leflunomide(LEF)
  LEF: Oral form, 20mg every other day for first 2 weeks then increasing to 20mg per day by the third week. Total treatment period is 16 weeks.
  Methotrexate:Off
  Arms: Leflunomide

SUMMARY:
In rheumatoid arthritis patients with active disease despite optimal treatment with methotrexate, the main objective of this pilot study is to use advance imaging tools such as magnetic resonance imaging and ultrasound to evaluate which treatment option is more efficacious: initiating methotrexate/sulfasalazine combination therapy, or switching to leflunomide monotherapy

ELIGIBILITY:
Inclusion Criteria

1. Male and female patients aged between 21 and 65 years.
2. Patients with no childbearing potential (For example postmenopausal or sterilised) or have decided not to have offspring(s).
3. All female patients must consent not to get pregnant/breastfeed, male patients must consent not to father a child and all must consent to practice effective birth control.
4. Fulfills either the 1987 ACR criteria and/or the 2010 ACR / EULAR RA Classification Criteria.
5. Seropositivity: Rheumatoid factor (RF) and/or anti -cyclic citrullinated protein antibodies (anti-CCP) must be positive.
6. MCPJ(s) and/or Wrist(s) joint(s) involvement.
7. Rheumatoid arthritis patients (less than 5 years duration) who remain at least moderately active based on DAS28 score of > 3.2, following 3 months of therapy with an optimal dose of methotrexate(e.g. at least 15 mg/week).
8. If patient is on oral corticosteroids, this should not exceeding 10mg prednisolone daily (or oral steroid equivalent) for at least 4 weeks and should be at an unchanged dose for at least 2 weeks before entering study.
9. If patient is on NSAIDs, this should be at an unchanged dose for at least 2 weeks before entering study.
10. Glomerular filtration rate > 60 mls/min/1.73m2.

Exclusion Criteria

1. Patient known to have the following medical condition(s) will be excluded:

   1. Other autoimmune disease /inflammatory joint disease/connective tissue disease ( e.g. lupus, seronegative spondylarthropathy (e.g. ankylosing spondylitis/psoriatic arthropathy ), reactive arthritis, overlap syndrome, primary sjogren syndrome and mixed connective tissue disease.)
   2. Inflammatory arthritis with onset before 18 years old.
   3. Current or previous history of cancer or lymphoproliferative disease.
   4. HIV positive status, Hepatitis B/C positive status.
   5. Persistent and/or severe infection in the previous 12 weeks.
   6. Major traumatic injury, terminal illness, or other medical condition(s)that could place the patient at risk to participate in the study.
   7. Clinically relevant cardiovascular (e.g unstable ischemic heart disease), neurological (e.g recent stroke), gastroenterology (e.g active peptic ulcer disease), renal (e.g chronic renal failure), hepatic (e.g alcoholic liver disease, fatty liver) and any other major systemic disease that could i) place the patient at risk to participate in the study; or ii) make protocol implementation difficult; or iii) make study results interpretation difficult.
   8. Presence of any known condition(s)/circumstance(s) which would negatively impact compliance or study completion.
2. Impaired laboratory parameters:

   1. Hemoglobin less than 10.5 g/dl, white blood count less than 4 x 10 (9)/L , platelet count less than 150 x 10(9)/L.
   2. Deranged Liver function test: e.g. elevated AST/ALT.
3. Wants to consume alcohol while taking the study medications.
4. Body weight that is less than 45 kg.
5. Pregnancy/Breastfeeding/Male patient wishing to father children.
6. Patients with the following medication history will be excluded:

   1. History of Glucose 6 Phosphate Dehydrogenase (G6PD) deficiency.
   2. Known allergy to: i) study medications; or ii) contrast; or iii) drugs whose chemical structures are similar (e.g. sulphonamides, salicylates, etc).
   3. On anticoagulation for any reasons.
   4. Previous treatment (within the last 4 weeks) with: i) oral corticosteroid greater than prednisolone equivalent of 10mg/day; or ii) parenteral/intra-articular corticosteroid injection.
   5. Previous treatment (within the last 12 weeks) with: i) other DMARDs such as sulfasalazine,hydroxychloroquine,chloroquine,gold salts, etc; or ii) investigational drug(s); or iii) other immunosuppressive agents such as cyclophosphamide,cyclosporin,azathioprine and any biologic agents, e.g. anti-TNF.
   6. Previous treatment(any duration) with i) Leflunomide; or ii) Sulfasalazine used together with methotrexate
7. Contraindication to MRI (e.g. pacemakers, metallic implants/stents, claustrophobia).

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2012-07; Primary Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
MRI synovitis score | four months

SECONDARY OUTCOMES:
MRI bone marrow edema score | 4 months
MRI erosion score | 4 months
US synovitis score | 4 months
clinical outcomes | 4 months
  Swollen/Tender joint counts, investigator's global assessment of disease activity (0-10), patient's assessment of disease activity (0-10), pain assessment by visual analogue scale (0-10), erythrocyte sedimentation rate, duration (mins) of early morning stiffness, and calculated disease activity indices

OTHER OUTCOMES:
US erosion score | 4 months
US tenosynovitis score | 4 months
MRI tenosynovitis score | 4 months
Adverse events | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: York Kiat Tan, MBBS,MRCP, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore, Singapore